CLINICAL TRIAL: NCT02543034
Title: Randomized, Controlled, Phase IV Study of Petrolatum Gauze, Allevyn, and New Dressing, Betafoam® in the Management of Split-Thickness Skin Graft Donor Site
Brief Title: Compare of Petrolatum Gauze, Allevyn, and New Dressing, Betafoam® in the Management of Split-Thickness Skin Graft Donor Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BTF14-KR-401
Record Dates: First submitted 2015-08-31; First posted 2015-09-07 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Skin Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Betafoam Wound Dressing (Experimental): This contains 3% povidone iodine. Dressing will be routinely changed on day 3 and day 7, and can be replaced anytime due to various factors such as exudate control, dislodgement, or by investigators' clinical decision.
  Interventions: Device: Betafoam Wound Dressing
- Petrolatum Gauze (Active Comparator): Dressing will be routinely changed on day 3 and day 7 and can be replaced anytime due to various factors such as exudate control, dislodgement, or by investigators' clinical decision.
  Interventions: Device: Petrolatum Gauze
- Allevyn Wound Dressing (Active Comparator): Allevyn adhesive wound dressing will be routinely changed on day 3 and day 7 and can be replaced anytime due to various factors such as exudate control, dislodgement, or by investigators' clinical decision.
  Interventions: Device: Allevyn Wound Dressing

INTERVENTIONS:
Device: Betafoam Wound Dressing — Foam dressing including Betadine iodine
  Other Names: Betafoam
  Arms: Betafoam Wound Dressing
Device: Petrolatum Gauze — Gauze dressing
  Arms: Petrolatum Gauze
Device: Allevyn Wound Dressing — Foam dressing
  Other Names: Allevyn
  Arms: Allevyn Wound Dressing

SUMMARY:
This study is a randomized, controlled, multi-centre, open-label, phase IV study.

Total 81 patients will be enrolled in this study. Patients will be randomly assigned to Betafoam®, petrolatum gauze or Allevyn for donor site wounds after skin graft operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who is same as or more than 19 years old
2. Patients who will receive elective skin harvest operation
3. Patients who is in lateral thigh or buttock with donor site area from 50 to 150 cm2
4. Female patients who use method of contraception for the study
5. Patients who voluntarily sign the informed consent

Exclusion Criteria:

1. Patients who are pregnant
2. Patients who are known to have allergy to the dressing product including PVPI
3. Known hyperthyroidism or other thyroid dysfunction such as nodular thyroid goiter, endemic goiter and Hashimoto's thyroiditis or patients who receive radioiodine therapy
4. Co-morbidities which may adversely affect wound healing for example a patient with uncontrolled diabetes (HbA1c > 8%), chronic renal failure, autoimmune disease, or immunocompromised patient
5. Patients who receive anticoagulants, steroids or immunosuppressants
6. Patients who have signs and symptoms of infection on enrollment and adversely affect wound healing
7. Patients who have skin lesion such as Herpes zoster on donor site
8. Burn of >20% total body surface area
9. If the donor site had been harvested on a previous occasion
10. Patients who is limited cognitive ability
11. Patients who are participating in or will plan to participate in other clinical trials
12. Other various conditions that the investigators judge inappropriate for enrolment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by speed of wound healing | 6 months
  Days needed for complete skin epithelialization in donor site wounds through routine swab culture (1 and 3 days) and visual assessment of wounds

SECONDARY OUTCOMES:
Efficacy as measured by adverse event collection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Lee, Dr., Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No